CLINICAL TRIAL: NCT04832165
Title: Effects of Inspiratory Muscle Training on Diaphragm Thickness, Inspiratory Muscle Pressure and Physical Function in Healthy Young Adults
Brief Title: Inspiratory Muscle Training on Diaphragm Thickness, Inspiratory Muscle Pressure and Physical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14/2021
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle inspiratory strength training (Experimental): An 8-week muscle inspiratory muscle strength training
  Interventions: Other: Inspiratory muscle strength training
- No training program (No Intervention): No intervention

INTERVENTIONS:
Other: Inspiratory muscle strength training — Inspiratory muscle training during 8 weeks, 30 inspirations at 60% of the PIM (maximum inspiratory pressure), 2 times a day for 5 days per week.
  Arms: Muscle inspiratory strength training

SUMMARY:
Fatigue of the respiratory muscles is one of the limitations of exercise at high intensity, although the mechanisms that explain it are not yet clear. This fatigue would cause a decrease in physical performance and could limit the functional capacity of the subject. In this sense, it has been shown that specific training of respiratory muscles, especially inspiratory muscles, improves their strength and resistance both in healthy people and in people with pathologies; managing to improve the quality of life and both physical and sports performance. This study, which follows the quantitative method and proposes an analytical, experimental, longitudinal and prospective design (with the aim of conducting a randomized clinical trial), proposes an intervention based on performing a specific training of inspiratory muscles for 8 weeks, taking 30 maximum inspirations at 60% of the PIM (maximum inspiratory pressure), 2 times a day for 5 days a week; with the aim of assessing the effects on inspiratory function, cardiorespiratory fitness when performing a stress test (Harvard step test) and diaphragm thickness measured by ultrasound. 40 healthy subjects between 18 and 25 years old will be recruited and divided into two groups: an experimental group (n = 20) and a control group (n = 20).

ELIGIBILITY:
Inclusion Criteria:

* healthy university students

Exclusion Criteria:

* Suffering or having suffered aortic aneurysm; pneumothorax; rib wall or pulmonary fistulas; recent trauma or surgery to the upper airway or thoracoabdominal; recent myocardial infarction or angina; retinal detachment, glaucoma, or recent eye surgery; increased intracranial pressure (tonsillar wedge, meningocele, hydrocephalus); abdominal hernias and acute middle ear problems.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Diaphragm muscle thickness | Change from baseline diaphragm muscle thickness at 8 weeks
  Diaphragm muscle thickness will be measured in mm by an ultrasound device

SECONDARY OUTCOMES:
Inspiratory muscle strength | Change from baseline inspiratory muscle strength at 8 weeks
  Inspiratory muscle strength will be measured in % by a POWER-breathe device
Physical Efficiency Index | Change from baseline physical efficiency index at 8 weeks
  Physical efficiency Index will be obtained by the Harvard Test

CONTACTS AND LOCATIONS:
Overall Officials: Berlanga, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No